CLINICAL TRIAL: NCT04715386
Title: Evaluation of Feasibility in the Prophylaxis of Radiation Dermatitis Severity in Cancer Patients
Brief Title: Feasibility in the Prophylaxis of Radiation Dermatitis Severity
Status: Terminated | Type: Observational
Why Stopped: slow accrual; investigator retired
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-007541; NCI-2023-00638 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2020-06-17; First posted 2021-01-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1- StrataXRT
  Interventions: Drug: StrataXRT

INTERVENTIONS:
Drug: StrataXRT — Patients will be asked to start topical application of their allocated topical preparation on the area of skin that will be irradiated at the onset of radiation therapy, every day until skin symptoms subside (see patient information pamphlet). Apply twice per day and can be reapplied as skin symptoms arise or as needed. The amount of StrataXRT provided to each patient will be recorded throughout treatment.

SUMMARY:
To compare radiation dermatitis severity in irradiated skin protected by an agent verses uncovered skin based on photographs and track patient reported outcomes with use of the agent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years
* Undergoing external beam radiotherapy for head/neck cancer at Mayo Clinic Rochester campus.

Note: patients undergoing concurrent chemotherapy are eligible.

* Able to provide informed written consent
* Willing to consent for photography of radiation field
* Receiving a dose ≥ 45 Gy and 20 fractions to both the area being treated and the area being used for comparison

Exclusion Criteria:

* Patients with active rash, pre-existing dermatitis, lupus, tattoos, scleroderma or other conditions within the treatment area that may make skin assessment for the study difficult per treating physician discretion.
* Patients with known allergic and other systemic skin diseases even if not directly affecting irradiated fields.
* Any medical condition that in the opinion of the investigator should exclude him/her from participating in the study.
* Enrolled in an investigational study where product was applied to the proposed study site within 30 days of the screening visit
* The skin area affected by radiation requires treatment with a concomitant medication or product (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with head and neck cancer
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
To compare radiation dermatitis severity in irradiated skin protected by an agent versus uncovered skin (internal control) based on photographs. | First day of treatment and last day of radiation therapy (approximately 6 weeks, but will vary per patient) +/- 4 days

SECONDARY OUTCOMES:
Patient reported outcomes | Upon study completion, on average 6 weeks, but will vary per patient
  Patients will be asked to complete a survey at the end of study that will ask them to provide feedback on the agent used during their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Petersen, MD, Principal Investigator — Mayo Clinic Radiation Oncology
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials